CLINICAL TRIAL: NCT01331681
Title: A Randomized, Double Masked, Active Controlled, Phase III Study of the Efficacy and Safety of Repeated Doses of Intravitreal VEGF Trap-Eye in Subjects With Diabetic Macular Edema
Brief Title: Intravitreal Aflibercept Injection in Vision Impairment Due to DME
Acronym: VIVID-DME
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 91745; 2010-022364-12 (EudraCT Number)
Record Dates: First submitted 2011-04-07; First posted 2011-04-08 (Estimated); Results first posted 2014-09-09 (Estimated); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus; Macular Edema
Keywords: Diabetic Macular Edema (DME); VEGF Trap-Eye; Best-corrected visual acuity (BCVA)
MeSH Terms: conditions — Diabetes Mellitus; Macular Edema | interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intravitreal Aflibercept Injection 2Q4 (Experimental): Participants received 2mg Intravitreal aflibercept injection (IAI) (EYLEA, VEGF Trap-Eye, BAY86-5321) every 4 weeks (2Q4).
  Interventions: Biological: VEGF Trap-Eye (BAY86-5321)
- Intravitreal Aflibercept Injection 2Q8 (Experimental): Participants received 2mg Intravitreal aflibercept injection (IAI) (EYLEA, VEGF Trap-Eye, BAY86-5321) every 4 weeks for 5 visits followed by injections every 8 weeks (2Q8).
  Interventions: Biological: VEGF Trap-Eye (BAY86-5321)
- Macular Laser Photocoagulation (Control) (Active Comparator): Participants received laser treatment at baseline and as needed at visits at which laser retreatment criteria were met, but no more frequently than every 12 weeks.
  Interventions: Procedure: Macular Laser Photocoagulation (Control)

INTERVENTIONS:
Biological: VEGF Trap-Eye (BAY86-5321) — Participants received 2mg Intravitreal aflibercept injection (IAI) (EYLEA, VEGF Trap-Eye, BAY86-5321) every 4 weeks (2Q4).
  Arms: Intravitreal Aflibercept Injection 2Q4
Biological: VEGF Trap-Eye (BAY86-5321) — Participants received 2mg Intravitreal aflibercept injection (IAI) (EYLEA, VEGF Trap-Eye, BAY86-5321) every 4 weeks for 5 visits followed by injections every 8 weeks (2Q8).
  Arms: Intravitreal Aflibercept Injection 2Q8
Procedure: Macular Laser Photocoagulation (Control) — Participants received laser treatment at baseline and as needed at visits at which laser retreatment criteria were met, but no more frequently than every 12 weeks.
  Arms: Macular Laser Photocoagulation (Control)

SUMMARY:
To determine the efficacy of intravitreally (IVT) administered VEGF Trap-Eye on the best-corrected visual acuity (BCVA) assessed by the early treatment diabetic retinopathy study (ETDRS) chart in subjects with diabetic macular edema (DME) with central involvement

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years with type 1 or 2 diabetes mellitus
* Subjects with DME secondary to diabetes mellitus involving the center of the macula in the study eye
* Decrease in vision determined to be primarily the result of DME in the study eye
* BCVA ETDRS letter score of 73 to 24 (20/40 to 20/320) in the study eye

Exclusion Criteria:

* Laser photocoagulation (panretinal or macular) in the study eye within 90 days of Day 1
* More than 2 previous macular laser treatments in the study eye
* Previous use of intraocular or periocular corticosteroids in the study eye within 120 days of Day 1
* Previous treatment with antiangiogenic drugs in either eye (pegaptanib sodium, bevacizumab, ranibizumab etc.) within 90 days of Day 1
* Active proliferative diabetic retinopathy (PDR) in the study eye, with the exception of inactive, regressed PDR
* Uncontrolled diabetes mellitus, as defined by HbA1c > 12%
* Only 1 functional eye even if that eye is otherwise eligible for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2011-05-09 (Actual); Primary Completion 2013-06-03 (Actual); Study Completion 2015-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (68):
- Australia (5):
  - Sydney, New South Wales
  - Westmead, New South Wales
  - East Melbourne, Victoria
  - Nedlands, Western Australia
  - Parramatta
- Austria (3):
  - Linz, Upper Austria
  - Linz
  - Vienna
- Czechia (4):
  - Faculty Hospital Hradec Kralove, Hradec Králové
  - Olomouc
  - Ostrava
  - Prague
- Denmark (2):
  - Århus C
  - Glostrup Municipality
- France (6):
  - Bordeaux
  - Créteil
  - Lyon
  - Nantes
  - Hopital Lariboisiere, Paris
  - Paris
- Germany (13):
  - Freiburg im Breisgau, Baden-Wurttemberg
  - Heidelberg, Baden-Wurttemberg
  - Tübingen, Baden-Wurttemberg
  - München, Bavaria
  - Darmstadt, Hesse
  - Göttingen, Lower Saxony
  - Aachen, North Rhine-Westphalia
  - Bonn, North Rhine-Westphalia
  - Cologne, North Rhine-Westphalia
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Mainz, Rhineland-Palatinate
  - Kiel, Schleswig-Holstein
  - Berlin
- Hungary (4):
  - Budapest
  - Debrecen
  - Veszprém
  - Zalaegerszeg
- Italy (5):
  - Rome, Lazio
  - Milan, Lombardy
  - Ancona, The Marches
  - Padua, Veneto
  - IRCCS Fondazione Ca' Granda Ospedale Maggiore Policlinico, Milan
- Japan (17):
  - Nagoya, Aichi-ken
  - Asahikwa, Hokkaido
  - Sapporo, Hokkaido
  - Kawasaki, Kanagawa
  - Sendai, Miyagi
  - Matsumoto, Nagano
  - Hirakata, Osaka
  - Chiyoda-ku, Tokyo
  - Itabashi-ku, Tokyo
  - Mitaka, Tokyo
  - Shinjuku-ku, Tokyo
  - Akita
  - Chiba
  - Fukuoka
  - Nagasaki
  - Osaka
  - Wakayama
- Poland (2):
  - Bytom
  - Wroclaw
- Spain (7):
  - Santiago de Compostela, A Coruña
  - San Cugat Del Vallès, Barcelona
  - Oviedo, Principality of Asturias
  - Alicante
  - Barcelona
  - Pamplona
  - Valencia

REFERENCES:
- [Background] Nanegrungsunk O, Gu SZ, Bressler SB, Du W, Amer F, Moini H, Bressler NM. Correlation of Change in Macular Thickness With Change in Visual Acuity in Diabetic Macular Edema: Post Hoc Analysis of VISTA and VIVID Trials. J Vitreoretin Dis. 2022 Jul 27;6(4):284-289. doi: 10.1177/24741264221099429. eCollection 2022 Jul-Aug. PMID 37007927
- [Background] Valentim CCS, Singh RP, Du W, Moini H, Talcott KE. Time to Resolution of Diabetic Macular Edema after Treatment with Intravitreal Aflibercept Injection or Laser in VISTA and VIVID. Ophthalmol Retina. 2023 Jan;7(1):24-32. doi: 10.1016/j.oret.2022.07.004. Epub 2022 Jul 14. PMID 35843487
- [Background] Dhoot DS, Moini H, Reed K, Du W, Vitti R, Berliner AJ, Singh RP. Functional outcomes of sustained improvement on Diabetic Retinopathy Severity Scale with intravitreal aflibercept in the VISTA and VIVID trials. Eye (Lond). 2023 Jul;37(10):2020-2025. doi: 10.1038/s41433-022-02058-7. Epub 2022 Apr 19. PMID 35440699
- [Result] Korobelnik JF, Do DV, Schmidt-Erfurth U, Boyer DS, Holz FG, Heier JS, Midena E, Kaiser PK, Terasaki H, Marcus DM, Nguyen QD, Jaffe GJ, Slakter JS, Simader C, Soo Y, Schmelter T, Yancopoulos GD, Stahl N, Vitti R, Berliner AJ, Zeitz O, Metzig C, Brown DM. Intravitreal aflibercept for diabetic macular edema. Ophthalmology. 2014 Nov;121(11):2247-54. doi: 10.1016/j.ophtha.2014.05.006. Epub 2014 Jul 8. PMID 25012934
- [Result] Brown DM, Schmidt-Erfurth U, Do DV, Holz FG, Boyer DS, Midena E, Heier JS, Terasaki H, Kaiser PK, Marcus DM, Nguyen QD, Jaffe GJ, Slakter JS, Simader C, Soo Y, Schmelter T, Yancopoulos GD, Stahl N, Vitti R, Berliner AJ, Zeitz O, Metzig C, Korobelnik JF. Intravitreal Aflibercept for Diabetic Macular Edema: 100-Week Results From the VISTA and VIVID Studies. Ophthalmology. 2015 Oct;122(10):2044-52. doi: 10.1016/j.ophtha.2015.06.017. Epub 2015 Jul 18. PMID 26198808
- [Result] Keating GM. Aflibercept: A Review of Its Use in Diabetic Macular Oedema. Drugs. 2015 Jul;75(10):1153-60. doi: 10.1007/s40265-015-0421-y. PMID 26056030
- [Result] Do DV, Gordon C, Suner IJ, Reed K, Moini H, Gibson A, Du W, Shah CP. Proliferative Diabetic Retinopathy Events in Patients With Diabetic Macular Edema: Post Hoc Analysis of VISTA and VIVID Trials. J Vitreoretin Dis. 2022 Jun 4;6(4):295-301. doi: 10.1177/24741264221093914. eCollection 2022 Jul-Aug. PMID 37007930
- [Derived] Dhoot DS, Moini H, Reed K, Silva FQ, Berliner A, Du W, Sharma S. INCIDENCE OF NEW DIABETIC MACULAR EDEMA IN FELLOW EYES OF PATIENTS IN THE VISTA AND VIVID STUDIES. Retina. 2023 Feb 1;43(2):254-262. doi: 10.1097/IAE.0000000000003658. Epub 2022 Oct 17. PMID 36265076
- [Derived] Midena E, Gillies M, Katz TA, Metzig C, Lu C, Ogura Y. Impact of Baseline Central Retinal Thickness on Outcomes in the VIVID-DME and VISTA-DME Studies. J Ophthalmol. 2018 Mar 29;2018:3640135. doi: 10.1155/2018/3640135. eCollection 2018. PMID 29785301
- [Derived] Staurenghi G, Feltgen N, Arnold JJ, Katz TA, Metzig C, Lu C, Holz FG; VIVID-DME and VISTA-DME study investigators. Impact of baseline Diabetic Retinopathy Severity Scale scores on visual outcomes in the VIVID-DME and VISTA-DME studies. Br J Ophthalmol. 2018 Jul;102(7):954-958. doi: 10.1136/bjophthalmol-2017-310664. Epub 2017 Oct 19. PMID 29051325
- [Derived] Wykoff CC, Marcus DM, Midena E, Korobelnik JF, Saroj N, Gibson A, Vitti R, Berliner AJ, Williams Liu Z, Zeitz O, Metzig C, Schmelter T, Heier JS. Intravitreal Aflibercept Injection in Eyes With Substantial Vision Loss After Laser Photocoagulation for Diabetic Macular Edema: Subanalysis of the VISTA and VIVID Randomized Clinical Trials. JAMA Ophthalmol. 2017 Feb 1;135(2):107-114. doi: 10.1001/jamaophthalmol.2016.4912. PMID 28006063
- [Derived] Ziemssen F, Schlottman PG, Lim JI, Agostini H, Lang GE, Bandello F. Initiation of intravitreal aflibercept injection treatment in patients with diabetic macular edema: a review of VIVID-DME and VISTA-DME data. Int J Retina Vitreous. 2016 Jul 11;2:16. doi: 10.1186/s40942-016-0041-z. eCollection 2016. PMID 27847634
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards — https://clinicaltrials.bayer.com/study/91745

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with diabetic macular edema (DME) secondary to diabetes mellitus involving the center of the macula in the study eye could participate in the study. The study was conducted at 73 study centers in Japan, European Countries and Australia between 09 May 2011(first participant first visit) and 30 Mar 2015 (last participant last visit).
Pre-assignment Details: Of 604 participants who were screened for inclusion in the study, 406 were randomized, and 404 received treatment.
Groups:
- Intravitreal Aflibercept Injection 2Q4: Participants received 2mg Intravitreal aflibercept injection (IAI) (EYLEA, VEGF [vascular endothelial growth factor] Trap-Eye, BAY86-5321) every 4 weeks (2Q4).
Period: Overall Study
Arm/Group | Intravitreal Aflibercept Injection 2Q4 | Intravitreal Aflibercept Injection 2Q8 | Macular Laser Photocoagulation (Control)
Started | 136 (randomized) | 135 (randomized) | 135 (randomized)
Participants Received Treatment | 136 (safety population) | 135 (safety population) | 133 (safety population)
Completed Week 52 | 125 | 121 | 115
Completed Week 100 | 115 | 110 | 105
Completed Week 148 | 101 | 101 | 100
Completed | 101 (Completed Week 148) | 101 (Completed Week 148) | 100 (Completed Week 148)
Not Completed | 35 | 34 | 35
Not completed — Adverse Event | 10 | 13 | 10
Not completed — Death | 6 | 6 | 2
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Withdrawal by Subject | 12 | 8 | 15
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Lost to Follow-up | 2 | 4 | 1
Not completed — Physician Decision | 2 | 0 | 4
Not completed — Therapeutic procedure required | 1 | 0 | 0
Not completed — Sponsor decision | 1 | 1 | 0
Not completed — Switching to other therapy | 0 | 0 | 1
Not completed — Not Received Study Treatment | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Control: Participants received laser treatment at baseline and as needed at visits at which laser retreatment criteria were met, but no more frequently than every 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Intravitreal Aflibercept Injection 2Q4 | Intravitreal Aflibercept Injection 2Q8 | Control | Total
Number analyzed (Participants) | 136 | 135 | 133 | 404
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.6 (8.6) | 64.2 (7.8) | 63.9 (8.6) | 63.6 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 47 | 54 | 154
  Male | 83 | 88 | 79 | 250

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in BCVA (Best Corrected Visual Acuity) as Measured by Early Treatment Diabetic Retinopathy Study (ETDRS) Letter Score at Week 52 - Last Observation Carried Forward (LOCF)
Description: Visual function of the study eye was assessed using the ETDRS protocol. A higher score represents better functioning.
Time Frame: Baseline up to Week 52
Population: Full analysis set (FAS) included all randomized participants who received any study treatment, had a baseline measurement of BCVA, and had at least 1 post-baseline assessment of BCVA.
Measure: Mean (Standard Deviation); unit: Letters correctly read
Arm/Group | Intravitreal Aflibercept Injection 2Q4 | Intravitreal Aflibercept Injection 2Q8 | Control
Number analyzed (Participants) | 136 | 135 | 132
Letters correctly read | 10.5 (9.55) | 10.7 (9.32) | 1.2 (10.65)
Statistical Analysis 1: Comparison: Intravitreal Aflibercept Injection 2Q4 vs Control; Hypothesis: Mean change identical in both groups; Test type: Superiority or Other; p < 0.0001, ANCOVA — Significance level alpha=0.025 for two sided test to adjust for multiplicity. Since this p-value was below the significance level of 0.025, the fixed sequence testing did continue with the first secondary endpoint; Treatment group and geographic region (Japan vs. Non-Japan) as factors and baseline value as covariate; Mean Difference (Final Values) = 9.3, 97.5% CI 2-sided [6.5 to 12.0] — Least square (LS) mean difference from ANCOVA. The estimate is calculated as EYLEA minus Laser. A positive value indicates a result in favor of EYLEA
Statistical Analysis 2: Comparison: Intravitreal Aflibercept Injection 2Q8 vs Control; Hypothesis: Mean change identical in both groups; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Treatment group and geographic region (Japan vs. Non-Japan) as factors and baseline value as covariate; Mean Difference (Final Values) = 9.1, 97.5% CI 2-sided [6.3 to 11.8] — LS mean difference from ANCOVA. The estimate is calculated as EYLEA minus Laser. A positive value indicates a result in favor of EYLEA

2. Secondary Outcome: Percentage of Participants Who Gained at Least 10 Letters in BCVA as Measured by ETDRS Letter Score Compared With Baseline at Week 52 - LOCF
Description: Visual function of the study eye was assessed using the ETDRS protocol. A higher score represents better functioning.
Time Frame: Baseline up to Week 52
Population: FAS.
Measure: Number; unit: Percentage of participants
Arm/Group | Intravitreal Aflibercept Injection 2Q4 | Intravitreal Aflibercept Injection 2Q8 | Control
Number analyzed (Participants) | 136 | 135 | 132
Percentage of participants | 54.4 | 53.3 | 25.8
Statistical Analysis 1: Comparison: Intravitreal Aflibercept Injection 2Q4 vs Control; Hypothesis: Probability to gain >= 10 letters identical in both groups; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Significance level alpha=0.025 for two sided test to adjust for multiplicity. Since this p-value and the preceding ones were below the significance level of 0.025, the fixed sequence testing did continue with the second secondary endpoint; Stratifying by geographic region (Japan vs non-Japan); CMH adjusted difference = 28.7, 97.5% CI 2-sided [15.8 to 41.6] — The estimate is calculated as EYLEA minus Laser. A positive value indicates a result in favor of EYLEA
Statistical Analysis 2: Comparison: Intravitreal Aflibercept Injection 2Q8 vs Control; Hypothesis: Probability to gain >= 10 letters identical in both groups; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Stratifying by geographic region (Japan vs non-Japan); CMH adjusted difference = 27.5, 97.5% CI 2-sided [14.6 to 40.5] — The estimate is calculated as EYLEA minus Laser. A positive value indicates a result in favor of EYLEA

3. Secondary Outcome: Percentage of Participants Who Gained at Least 15 Letters in BCVA as Measured by ETDRS Letter Score Compared With Baseline at Week 52 - LOCF
Description: Visual function of the study eye was assessed using the ETDRS protocol. A higher score represents better functioning.
Time Frame: Baseline up to Week 52
Population: FAS.
Measure: Number; unit: Percentage of participants
Arm/Group | Intravitreal Aflibercept Injection 2Q4 | Intravitreal Aflibercept Injection 2Q8 | Control
Number analyzed (Participants) | 136 | 135 | 132
Percentage of participants | 32.4 | 33.3 | 9.1
Statistical Analysis 1: Comparison: Intravitreal Aflibercept Injection 2Q4 vs Control; Hypothesis: Probability to gain >= 15 letters identical in both groups; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Significance level alpha=0.025 for two sided test to adjust for multiplicity. Since this p-value and the preceding ones were below the significance level of 0.025, the fixed sequence testing did continue with the third secondary endpoint; Stratifying by geographic region (Japan vs non-Japan); CMH adjusted difference = 23.3, 97.5% CI 2-sided [12.6 to 33.9] — The estimate is calculated as EYLEA minus Laser. A positive value indicates a result in favor of EYLEA
Statistical Analysis 2: Comparison: Intravitreal Aflibercept Injection 2Q8 vs Control; Hypothesis: Probability to gain >= 15 letters identical in both groups; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Stratifying by geographic region (Japan vs non-Japan); CMH adjusted difference = 24.2, 97.5% CI 2-sided [13.5 to 34.9] — The estimate is calculated as EYLEA minus Laser. A positive value indicates a result in favor of EYLEA

4. Secondary Outcome: Percentage of Participants With a ≥2-step Improvement From Baseline in the ETDRS DRSS (Diabetic Retinopathy Severity Score) as Assessed by FP (Fundus Photography) at Week 52 - LOCF
Description: Baseline ETDRS DRSS: None (level 10); Mild to moderate nonproliferative DR (levels 14, 15, 20, 35, and 43); Moderately severe/severe nonproliferative DR (levels 47 and 53); Mild/moderate/high-risk/advanced proliferative DR (levels 61, 65, 71,75, 81, and 85)
Time Frame: Baseline up to Week 52
Population: Full-Analysis Set with assessment for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Intravitreal Aflibercept Injection 2Q4 | Intravitreal Aflibercept Injection 2Q8 | Control
Number analyzed (Participants) | 81 | 83 | 80
Percentage of participants | 33.3 | 27.7 | 7.5
Statistical Analysis 1: Comparison: Intravitreal Aflibercept Injection 2Q4 vs Control; Hypothesis: Probability to improve by >= 2 steps identical in both groups; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Significance level alpha=0.025 for two sided test to adjust for multiplicity. Since this p-value and the preceding ones were below the significance level of 0.025, the fixed sequence testing did continue with the fourth secondary endpoint; Stratifying by geographic region (Japan vs non-Japan); CMH adjusted difference = 25.8, 97.5% CI 2-sided [12.2 to 39.4] — The estimate is calculated as EYLEA minus Laser. A positive value indicates a result in favor of EYLEA
Statistical Analysis 2: Comparison: Intravitreal Aflibercept Injection 2Q8 vs Control; Hypothesis: Probability to improve by >= 2 steps identical in both groups; Test type: Superiority or Other; p = 0.0006, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; Stratifying by geographic region (Japan vs non-Japan); CMH adjusted difference = 19.3, 97.5% CI 2-sided [6.6 to 32.1] — The estimate is calculated as EYLEA minus Laser. A positive value indicates a result in favor of EYLEA

5. Secondary Outcome: Change From Baseline in Central Retinal Thickness (CRT) at Week 52 as Assessed on Optical Coherence Tomography (OCT) - LOCF
Time Frame: Baseline up to Week 52
Population: Full-Analysis Set with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | Intravitreal Aflibercept Injection 2Q4 | Intravitreal Aflibercept Injection 2Q8 | Control
Number analyzed (Participants) | 135 | 135 | 132
micrometer | -195.0 (146.59) | -192.4 (149.89) | -66.2 (138.99)
Statistical Analysis 1: Comparison: Intravitreal Aflibercept Injection 2Q4 vs Control; Hypothesis: Mean change identical in both groups; Test type: Superiority or Other; p < 0.0001, ANCOVA — Significance level alpha=0.025 for two sided test to adjust for multiplicity. Since this p-value and the preceding ones were below the significance level of 0.025, the fixed sequence testing did continue with the fifth secondary endpoint; Treatment group and geographic region (Japan vs. Non-Japan) as factors and baseline value as covariate; Mean Difference (Final Values) = -157.0, 97.5% CI 2-sided [-190.9 to -123.1] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Intravitreal Aflibercept Injection 2Q8 vs Control; Hypothesis: Mean change identical in both groups; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 5, analysis 1]; Treatment group and geographic region (Japan vs. Non-Japan) as factors and baseline value as covariate; Mean Difference (Final Values) = -142.8, 97.5% CI 2-sided [-179.3 to -106.3] — LS mean difference from ANCOVA. The estimate is calculated as EYLEA minus Laser. A negative value indicates a result in favor of EYLEA

6. Secondary Outcome: Change From Baseline in National Eye Institute 25-item Visual Function Questionnaire (NEI VFQ-25) Near Activities Subscale at Week 52 - LOCF
Description: The NEI VFQ-25 total score ranges from 0-100 with a score of 0 being the worst outcome and 100 being the best outcome. The NEI VFQ questionnaire is organized as a collection of subscales that are all scored from 0-100. Near activities are defined as reading ordinary print in newspapers, performing work or hobbies requiring near vision, or finding something on a crowded shelf.
Time Frame: Baseline up to Week 52
Population: Full-Analysis Set with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Intravitreal Aflibercept Injection 2Q4 | Intravitreal Aflibercept Injection 2Q8 | Control
Number analyzed (Participants) | 128 | 134 | 120
Scores on a scale | 5.73 (18.932) | 5.29 (19.058) | 3.54 (16.768)
Statistical Analysis 1: Comparison: Intravitreal Aflibercept Injection 2Q4 vs Control; Hypothesis: Mean change identical in both groups; Test type: Superiority or Other; p = 0.2208, ANCOVA — Significance level alpha=0.025 for two sided test to adjust for multiplicity. Since this p-value is not below of 0.025, the fixed sequence testing stops here. The sixth secondary endpoint cannot be tested confirmatory; Treatment group and geographic region (Japan vs. Non-Japan) as factors and baseline value as covariate; Mean Difference (Final Values) = 2.41, 97.5% CI 2-sided [-2.01 to 6.82] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Intravitreal Aflibercept Injection 2Q8 vs Control; Hypothesis: Mean change identical in both groups; Test type: Superiority or Other; p = 0.5537, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Treatment group and geographic region (Japan vs. Non-Japan) as factors and baseline value as covariate; Mean Difference (Final Values) = -1.21, 97.5% CI 2-sided [-5.79 to 3.37] — [estimate comment as in outcome 1, analysis 2]

7. Secondary Outcome: Change From Baseline in National Eye Institute 25-item Visual Function Questionnaire (NEI VFQ-25) Distance Activities Subscale at Week 52 - LOCF
Description: The NEI VFQ-25 total score ranges from 0-100 with a score of 0 being the worst outcome and 100 being the best outcome. The NEI VFQ questionnaire is organized as a collection of subscales that are all scored from 0-100. Distance activities are defined as reading street signs or names on stores, and going down stairs, steps, or curbs.
Time Frame: Baseline up to Week 52
Population: Full-Analysis Set with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Intravitreal Aflibercept Injection 2Q4 | Intravitreal Aflibercept Injection 2Q8 | Control
Number analyzed (Participants) | 128 | 134 | 120
Scores on a scale | 0.94 (16.487) | 5.32 (18.475) | 2.26 (15.923)
Statistical Analysis 1: Comparison: Intravitreal Aflibercept Injection 2Q4 vs Control; Hypothesis: Mean change identical in both groups; Test type: Superiority or Other; p = 0.5138, ANCOVA; Mean Difference (Final Values) = -1.19, 97.5% CI 2-sided [-5.29 to 2.91] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Intravitreal Aflibercept Injection 2Q8 vs Control; Hypothesis: Mean change identical in both groups; Test type: Superiority or Other; p = 0.8498, ANCOVA; Mean Difference (Final Values) = -0.37, 97.5% CI 2-sided [-4.79 to 4.05] — [estimate comment as in outcome 1, analysis 2]

ADVERSE EVENTS:
Time Frame: For each subject from his first study drug injection until 30 days after the last study drug injection at the latest up to termination visit at Week 148
Groups:
- Macular Laser Photocoagulation (Control): Participants received laser treatment at baseline and as needed at visits at which laser retreatment criteria were met, but no more frequently than every 12 weeks. During year 3 laser patients could receive IAI as needed (PRN) .
Arm/Group | Intravitreal Aflibercept Injection 2Q4 | Intravitreal Aflibercept Injection 2Q8 | Macular Laser Photocoagulation (Control)
Serious Adverse Events (participants affected / at risk) | 63 | 60 | 51
Other Adverse Events (participants affected / at risk) | 117/136 | 122/135 | 113/133
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Intravitreal Aflibercept Injection 2Q4 | Intravitreal Aflibercept Injection 2Q8 | Macular Laser Photocoagulation (Control)
Anaemia (Blood and lymphatic system disorders) | 0/136 (0) | 1/135 (1) | 1/133 (1)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1/136 (2) | 0/135 (0) | 0/133 (0)
Neutropenia (Blood and lymphatic system disorders) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Acute coronary syndrome (Cardiac disorders) | 0/136 (0) | 0/135 (0) | 1/133 (1)
Acute myocardial infarction (Cardiac disorders) | 2/136 (2) | 0/135 (0) | 3/133 (3)
Angina unstable (Cardiac disorders) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Arrhythmia (Cardiac disorders) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Atrioventricular block complete (Cardiac disorders) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Bundle branch block right (Cardiac disorders) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Cardiac disorder (Cardiac disorders) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Cardiac failure (Cardiac disorders) | 1/136 (1) | 2/135 (2) | 2/133 (2)
Cardiac failure acute (Cardiac disorders) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Cardiac failure chronic (Cardiac disorders) | 0/136 (0) | 0/135 (0) | 1/133 (2)
Cardiac failure congestive (Cardiac disorders) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Cardiac sarcoidosis (Cardiac disorders) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Cardiac valve disease (Cardiac disorders) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Cardiogenic shock (Cardiac disorders) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Coronary artery disease (Cardiac disorders) | 2/136 (3) | 0/135 (0) | 1/133 (1)
Coronary artery stenosis (Cardiac disorders) | 2/136 (2) | 0/135 (0) | 0/133 (0)
Hypertensive heart disease (Cardiac disorders) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 0/136 (0) | 0/135 (0) | 1/133 (1)
Left ventricular failure (Cardiac disorders) | 1/136 (2) | 0/135 (0) | 0/133 (0)
Mitral valve stenosis (Cardiac disorders) | 0/136 (0) | 0/135 (0) | 1/133 (1)
Myocardial infarction (Cardiac disorders) | 4/136 (4) | 1/135 (1) | 1/133 (1)
Myocardial ischaemia (Cardiac disorders) | 1/136 (1) | 0/135 (0) | 1/133 (1)
Ventricular arrhythmia (Cardiac disorders) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Ventricular tachycardia (Cardiac disorders) | 1/136 (2) | 0/135 (0) | 0/133 (0)
Deafness (Ear and labyrinth disorders) | 0/136 (0) | 0/135 (0) | 1/133 (1)
Vertigo (Ear and labyrinth disorders) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Toxic nodular goitre (Endocrine disorders) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Cataract (Eye disorders) | 5/136 (8) | 7/135 (11) | 2/133 (2)
Cataract subcapsular (Eye disorders) | 1/136 (1) | 2/135 (2) | 0/133 (0)
Diabetic retinopathy (Eye disorders) | 0/136 (0) | 0/135 (0) | 2/133 (2)
Iridocyclitis (Eye disorders) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Macular degeneration (Eye disorders) | 0/136 (0) | 0/135 (0) | 1/133 (1)
Macular fibrosis (Eye disorders) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Macular hole (Eye disorders) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Optic atrophy (Eye disorders) | 0/136 (0) | 0/135 (0) | 1/133 (1)
Posterior capsule opacification (Eye disorders) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Retinal artery occlusion (Eye disorders) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Retinal detachment (Eye disorders) | 0/136 (0) | 2/135 (2) | 1/133 (1)
Retinal exudates (Eye disorders) | 0/136 (0) | 0/135 (0) | 1/133 (1)
Retinal neovascularisation (Eye disorders) | 1/136 (1) | 0/135 (0) | 3/133 (4)
Retinal vascular disorder (Eye disorders) | 0/136 (0) | 0/135 (0) | 1/133 (2)
Retinopathy proliferative (Eye disorders) | 0/136 (0) | 0/135 (0) | 1/133 (1)
Vitreous haemorrhage (Eye disorders) | 4/136 (5) | 1/135 (1) | 2/133 (4)
Abdominal pain upper (Gastrointestinal disorders) | 1/136 (1) | 1/135 (1) | 0/133 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Enterocolitis (Gastrointestinal disorders) | 0/136 (0) | 0/135 (0) | 1/133 (1)
Gastric ulcer (Gastrointestinal disorders) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Ileus (Gastrointestinal disorders) | 0/136 (0) | 2/135 (2) | 0/133 (0)
Inguinal hernia (Gastrointestinal disorders) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Reflux gastritis (Gastrointestinal disorders) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Chest pain (General disorders) | 0/136 (0) | 0/135 (0) | 1/133 (1)
Death (General disorders) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Device failure (General disorders) | 0/136 (0) | 0/135 (0) | 1/133 (2)
Generalised oedema (General disorders) | 0/136 (0) | 1/135 (2) | 0/133 (0)
Injection site injury (General disorders) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Oedema peripheral (General disorders) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Cholecystitis (Hepatobiliary disorders) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Cholelithiasis (Hepatobiliary disorders) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Cellulitis (Infections and infestations) | 0/136 (0) | 2/135 (2) | 2/133 (2)
Cholecystitis infective (Infections and infestations) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Endophthalmitis (Infections and infestations) | 1/136 (1) | 0/135 (0) | 1/133 (1)
Gangrene (Infections and infestations) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Gastroenteritis (Infections and infestations) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Infected dermal cyst (Infections and infestations) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Infected skin ulcer (Infections and infestations) | 0/136 (0) | 0/135 (0) | 1/133 (1)
Osteomyelitis (Infections and infestations) | 0/136 (0) | 0/135 (0) | 1/133 (1)
Pilonidal cyst (Infections and infestations) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Pneumonia (Infections and infestations) | 1/136 (1) | 3/135 (3) | 0/133 (0)
Pyelonephritis (Infections and infestations) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Salmonellosis (Infections and infestations) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Sepsis (Infections and infestations) | 0/136 (0) | 1/135 (1) | 1/133 (1)
Urinary tract infection (Infections and infestations) | 0/136 (0) | 0/135 (0) | 1/133 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Brain contusion (Injury, poisoning and procedural complications) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Brain herniation (Injury, poisoning and procedural complications) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0/136 (0) | 0/135 (0) | 1/133 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Fracture (Injury, poisoning and procedural complications) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Head injury (Injury, poisoning and procedural complications) | 0/136 (0) | 0/135 (0) | 1/133 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 3/136 (3) | 1/135 (1) | 0/133 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0/136 (0) | 0/135 (0) | 1/133 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1/136 (1) | 0/135 (0) | 1/133 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Traumatic arthrosis (Injury, poisoning and procedural complications) | 1/136 (2) | 0/135 (0) | 0/133 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 0/136 (0) | 0/135 (0) | 1/133 (1)
Catheterisation cardiac (Investigations) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Electrocardiogram ST segment depression (Investigations) | 0/136 (0) | 0/135 (0) | 1/133 (1)
Visual acuity tests abnormal (Investigations) | 0/136 (0) | 0/135 (0) | 1/133 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1/136 (2) | 2/135 (2) | 1/133 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Fluid retention (Metabolism and nutrition disorders) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0/136 (0) | 2/135 (2) | 2/133 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0/136 (0) | 0/135 (0) | 1/133 (1)
Ketoacidosis (Metabolism and nutrition disorders) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1/136 (2) | 0/135 (0) | 0/133 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1/136 (1) | 0/135 (0) | 1/133 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0/136 (0) | 0/135 (0) | 2/133 (2)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0/136 (0) | 0/135 (0) | 1/133 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2/136 (2) | 0/135 (0) | 0/133 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0/136 (0) | 1/135 (1) | 1/133 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0/136 (0) | 1/135 (2) | 0/133 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0/136 (0) | 0/135 (0) | 1/133 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0/136 (0) | 0/135 (0) | 1/133 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 0/136 (0) | 0/135 (0) | 1/133 (1)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Anaplastic astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/136 (0) | 1/135 (1) | 0/133 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/136 (1) | 0/135 (0) | 1/133 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/136 (1) | 0/135 (0) | 1/133 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/136 (1) | 1/135 (1) | 0/133 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/136 (0) | 1/135 (1) | 1/133 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/136 (0) | 1/135 (1) | 1/133 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Pancreatic carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Prostate cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/136 (2) | 0/135 (0) | 1/133 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Brain stem infarction (Nervous system disorders) | 0/136 (0) | 0/135 (0) | 1/133 (1)
Cauda equina syndrome (Nervous system disorders) | 0/136 (0) | 0/135 (0) | 1/133 (1)
Cerebral atrophy (Nervous system disorders) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Cerebral haematoma (Nervous system disorders) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Cerebral haemorrhage (Nervous system disorders) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Cerebrovascular accident (Nervous system disorders) | 4/136 (4) | 1/135 (1) | 1/133 (1)
Ischaemic stroke (Nervous system disorders) | 2/136 (2) | 0/135 (0) | 1/133 (1)
Loss of consciousness (Nervous system disorders) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Nerve compression (Nervous system disorders) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Syncope (Nervous system disorders) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Depression (Psychiatric disorders) | 0/136 (0) | 0/135 (0) | 1/133 (2)
Suicide attempt (Psychiatric disorders) | 0/136 (0) | 0/135 (0) | 1/133 (1)
Acute kidney injury (Renal and urinary disorders) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Chronic kidney disease (Renal and urinary disorders) | 1/136 (1) | 1/135 (1) | 0/133 (0)
Nephrolithiasis (Renal and urinary disorders) | 0/136 (0) | 0/135 (0) | 1/133 (1)
Renal artery stenosis (Renal and urinary disorders) | 1/136 (1) | 0/135 (0) | 1/133 (1)
Renal failure (Renal and urinary disorders) | 1/136 (1) | 2/135 (2) | 0/133 (0)
Renal impairment (Renal and urinary disorders) | 0/136 (0) | 1/135 (2) | 0/133 (0)
Stress urinary incontinence (Renal and urinary disorders) | 0/136 (0) | 0/135 (0) | 1/133 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/136 (0) | 1/135 (1) | 2/133 (2)
Uterine polyp (Reproductive system and breast disorders) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0/136 (0) | 0/135 (0) | 1/133 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0/136 (0) | 0/135 (0) | 1/133 (1)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1/136 (1) | 1/135 (1) | 0/133 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1/136 (2) | 0/135 (0) | 2/133 (2)
Psoriasis (Skin and subcutaneous tissue disorders) | 0/136 (0) | 0/135 (0) | 2/133 (3)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0/136 (0) | 1/135 (1) | 2/133 (2)
Arteriovenous shunt operation (Surgical and medical procedures) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Cataract operation (Surgical and medical procedures) | 3/136 (3) | 1/135 (1) | 2/133 (3)
Hip arthroplasty (Surgical and medical procedures) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Osteosynthesis (Surgical and medical procedures) | 0/136 (0) | 0/135 (0) | 1/133 (1)
Peripheral artery bypass (Surgical and medical procedures) | 1/136 (1) | 0/135 (0) | 1/133 (1)
Radical prostatectomy (Surgical and medical procedures) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Transurethral prostatectomy (Surgical and medical procedures) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Vitrectomy (Surgical and medical procedures) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Arterial haemorrhage (Vascular disorders) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Arteriosclerosis (Vascular disorders) | 0/136 (0) | 1/135 (1) | 0/133 (0)
Circulatory collapse (Vascular disorders) | 0/136 (0) | 0/135 (0) | 1/133 (1)
Deep vein thrombosis (Vascular disorders) | 1/136 (1) | 0/135 (0) | 0/133 (0)
Hypertension (Vascular disorders) | 1/136 (1) | 1/135 (1) | 0/133 (0)
Lymphoedema (Vascular disorders) | 0/136 (0) | 0/135 (0) | 1/133 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1/136 (1) | 2/135 (2) | 3/133 (3)
Peripheral artery stenosis (Vascular disorders) | 1/136 (1) | 0/135 (0) | 1/133 (1)
Peripheral ischaemia (Vascular disorders) | 0/136 (0) | 1/135 (1) | 1/133 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravitreal Aflibercept Injection 2Q4 (N=136) | Intravitreal Aflibercept Injection 2Q8 (N=135) | Macular Laser Photocoagulation (Control) (N=133)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 3 (3) | 8 (8)
Cataract (Eye disorders) | 31 (43) | 26 (37) | 17 (29)
Cataract cortical (Eye disorders) | 7 (12) | 6 (7) | 1 (3)
Cataract subcapsular (Eye disorders) | 11 (16) | 5 (6) | 4 (4)
Conjunctival haemorrhage (Eye disorders) | 43 (59) | 39 (58) | 17 (26)
Conjunctival hyperaemia (Eye disorders) | 8 (10) | 3 (5) | 9 (15)
Corneal erosion (Eye disorders) | 9 (11) | 8 (10) | 7 (16)
Cystoid macular oedema (Eye disorders) | 10 (18) | 20 (67) | 18 (51)
Diabetic retinal oedema (Eye disorders) | 33 (49) | 23 (44) | 18 (25)
Eye pain (Eye disorders) | 15 (34) | 10 (19) | 10 (15)
Macular fibrosis (Eye disorders) | 10 (13) | 12 (17) | 11 (14)
Macular oedema (Eye disorders) | 21 (41) | 20 (31) | 22 (46)
Ocular hyperaemia (Eye disorders) | 5 (12) | 7 (9) | 4 (5)
Ocular hypertension (Eye disorders) | 10 (21) | 4 (9) | 6 (7)
Posterior capsule opacification (Eye disorders) | 10 (15) | 12 (15) | 10 (18)
Punctate keratitis (Eye disorders) | 7 (13) | 11 (19) | 8 (14)
Retinal aneurysm (Eye disorders) | 14 (26) | 12 (26) | 9 (16)
Retinal exudates (Eye disorders) | 20 (38) | 22 (49) | 15 (32)
Retinal haemorrhage (Eye disorders) | 21 (35) | 25 (64) | 21 (63)
Retinal vascular disorder (Eye disorders) | 9 (20) | 8 (13) | 5 (10)
Visual acuity reduced (Eye disorders) | 33 (64) | 33 (81) | 30 (57)
Vitreous detachment (Eye disorders) | 9 (12) | 10 (11) | 5 (7)
Vitreous floaters (Eye disorders) | 13 (14) | 5 (7) | 4 (4)
Vitreous haemorrhage (Eye disorders) | 7 (14) | 11 (11) | 8 (12)
Bronchitis (Infections and infestations) | 12 (16) | 5 (5) | 9 (10)
Conjunctivitis (Infections and infestations) | 14 (16) | 13 (20) | 8 (10)
Influenza (Infections and infestations) | 7 (10) | 11 (11) | 13 (16)
Nasopharyngitis (Infections and infestations) | 38 (67) | 39 (69) | 34 (62)
Urinary tract infection (Infections and infestations) | 6 (8) | 11 (22) | 6 (11)
Blood creatinine increased (Investigations) | 7 (8) | 6 (6) | 5 (5)
Blood glucose increased (Investigations) | 10 (13) | 7 (8) | 8 (10)
Blood urea increased (Investigations) | 6 (8) | 10 (10) | 6 (7)
Glycosylated haemoglobin increased (Investigations) | 12 (15) | 11 (12) | 11 (11)
Intraocular pressure increased (Investigations) | 28 (77) | 18 (51) | 16 (32)
Visual acuity tests abnormal (Investigations) | 19 (35) | 22 (63) | 32 (49)
Diabetes mellitus (Metabolism and nutrition disorders) | 6 (6) | 10 (12) | 9 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (3) | 11 (11)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 9 (9) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 6 (6) | 7 (10)
Hypertension (Vascular disorders) | 23 (32) | 25 (37) | 24 (41)
Dry eye (Eye disorders) | 5 (9) | 5 (7) | 8 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CONTRACT PARTNERS shall provide to BSP (Bayer Schering Pharma) any proposed publication or oral at least sixty (60) days prior to the intended submission or presentation. If BSP does not notify CONTRACT PARTNERS within sixty (60) days of BSP's receipt of the intended PUBLICATION, CONTRACT PARTNERS shall be free to publish. CONTRACT PARTNERS acknowledge that in case of multi-centre studies the RESULTS of the STUDY are to be published only through coordination by Bayer.